CLINICAL TRIAL: NCT00359619
Title: A Long-term, Follow-up of the Immunogenicity and Safety of GlaxoSmithKline Biologicals' Novel HPV Vaccine in Healthy Female Subjects Vaccinated in the Primary Study
Brief Title: Human Papillomavirus Vaccine Immunogenicity and Safety Trial in Young Adult Women With GSK Biologicals Novel HPV Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108052 (FU month 18); 107919 (Other: GSK); 107921 (Other: GSK); 107918 (Other: GSK); 2004-003766-14 (EudraCT Number); NCT00359502 (obsolete NCT alias); NCT00359528 (obsolete NCT alias); NCT00359827 (obsolete NCT alias)
Record Dates: First submitted 2006-07-18; First posted 2006-08-02 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus; Papillomavirus Vaccines
Keywords: HPV vaccine
MeSH Terms: conditions — Papillomavirus Infections

ARMS (7):
- Cervarix Group (Active Comparator): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: CervarixTM
- Cervarix 1 Group (Experimental): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine formulation 1 at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: HPV investigational vaccine GSK568893A, different formulations
- Cervarix 2 Group (Experimental): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine formulation 2 at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: HPV investigational vaccine GSK568893A, different formulations
- Cervarix 3 Group (Experimental): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine formulation 3 at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: HPV investigational vaccine GSK568893A, different formulations
- Cervarix 4 Group (Experimental): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine formulation 4 at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: HPV investigational vaccine GSK568893A, different formulations
- Cervarix 5 Group (Experimental): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine formulation 5 at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: HPV investigational vaccine GSK568893A, different formulations
- Cervarix 6 Group (Experimental): Female subjects, aged 18 to 25 years at the time of first vaccination, received 3 doses of Cervarix vaccine formulation 6 at Months 0, 1 and 6. The vaccine was administered intramuscularly into the deltoid region of the non-dominant arm.
  Interventions: Biological: HPV investigational vaccine GSK568893A, different formulations

INTERVENTIONS:
Biological: CervarixTM — Subjects were administered three doses of HPV vaccine
  Arms: Cervarix Group
Biological: HPV investigational vaccine GSK568893A, different formulations — Subjects were administered three doses of HPV investigational vaccine
  Arms: Cervarix 1 Group; Cervarix 2 Group; Cervarix 3 Group; Cervarix 4 Group; Cervarix 5 Group; Cervarix 6 Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Indeed, certain oncogenic types of HPV can infect the cervix (part of the uterus or womb). This infection may go away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. GlaxoSmithKline Biological's has developed a HPV vaccine against the oncogenic types HPV-16 and HPV-18 formulated with the AS04 adjuvant (control vaccine) and is also evaluating novel HPV vaccines formulations. This study will evaluate the long-term immunogenicity and safety of a novel GSK Biological's vaccine in approximately 376 subjects who received the novel vaccine or the control vaccine administered in the primary study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A female who enrolled in the study 102115 and received three doses of vaccine.
* Written informed consent obtained from the subject prior to enrolment.

Exclusion Criteria:

* Use (or planned use during the study period) of any investigational or non-registered product or off-label use of licensed product (drug or vaccine).
* Chronic administration of immunosuppressants or other immune-modifying drugs occurring less than three months prior to blood sampling.
* Administration of immunoglobulins and/or any blood products within the three months preceding blood sampling.
* Planned administration of any HPV vaccine, other than that foreseen by the study protocol, during the study period.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 383 (Actual)
Dates: Start 2006-09-12 (Actual); Primary Completion 2007-01-30 (Actual); Study Completion 2007-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (3):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Salt Lake City, Utah
- Belgium (6):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Tienen
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=1524

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 108052 (FU month 18) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108052 (FU month 18) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108052 (FU month 18) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 108052 (FU month 18) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108052 (FU month 18) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is a safety follow-up of the primary study NCT00231413, starting from Month 18 post-vaccination.
Pre-assignment Details: A total number of 383 subjects were enrolled in the primary study. A total of 193, 216, 182 and 166 subjects attended Month 18, Month 24, Month 36 and Month 48 visits, respectively. No separate demography data was tabulated for these intermediate timepoints, as statistics were computed only after the last study visit at Month 48.
Period: Overall Study
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Started | 88 | 50 | 49 | 48 | 48 | 50 | 50
Completed | 80 | 45 | 42 | 45 | 45 | 45 | 46
Not Completed | 8 | 5 | 7 | 3 | 3 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 4 | 2 | 2 | 0 | 3
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 2 | 1 | 1 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group | Total
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50 | 383
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.9 (2.03) | 21.5 (2.18) | 21.2 (2.07) | 21.1 (2.09) | 21.4 (2.27) | 21.2 (2.26) | 20.7 (1.91) | 21.1 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 50 | 49 | 48 | 48 | 50 | 50 | 383
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus-16 (HPV-16) Antibodies.
Description: Seroconversion was defined as the appearance of antibodies in the serum of subjects seronegative before vaccination. Seronegative subjects are subjects who had an antibody concentration below cut-off value. The assessed cut-off value was 8 ELISA units per milliliter (EL.U/mL).
Time Frame: At Months 18, 24, 36 and 48.
Population: The analysis was performed on the According-to-Protocol cohort for Immunogenicity, which included all evaluable subjects for whom immunogenicity data were available, and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 28 | 12 | 11 | 9 | 16 | 15 | 15
subjects
  Anti-HPV-16, Month 18 (N=27,10,9,8,14,13,13) | 27 | 10 | 9 | 8 | 14 | 13 | 13
  Anti-HPV-16, Month 24 (N=28,12,11,9,16,15,15) | 28 | 12 | 11 | 9 | 16 | 15 | 15
  Anti-HPV-16, Month 36 (N=28,12,11,9,16,15,15) | 28 | 12 | 11 | 9 | 16 | 15 | 15
  Anti-HPV-16, Month 48 (N=28,12,11,9,16,15,15) | 28 | 12 | 11 | 9 | 16 | 15 | 15

2. Primary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus-16 (HPV-16) Antibodies.
Description: Antibody titers were expressed as GMTs. The reference cut-off value was greater than or equal to (≥) 8 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 28 | 12 | 11 | 9 | 16 | 15 | 15
EL.U/mL
  Anti-HPV-16 Month 18 (N=27,10,9,8,14,13,13) | 1933.9 [1318.0 to 2837.5] | 1868.3 [1263.0 to 2763.8] | 1902.3 [603.5 to 5996.7] | 1996.4 [1017.8 to 3915.8] | 1437.1 [777.3 to 2657.0] | 2200.3 [1284.4 to 3769.4] | 1769.8 [914.9 to 3423.7]
  Anti-HPV-16 Month 24 (N=28,12,11,9,16,15,15) | 1477.1 [1039.3 to 2099.3] | 1381.6 [942.1 to 2026.4] | 1339.9 [553.1 to 3246.1] | 1520.6 [916.6 to 2522.5] | 1264.4 [718.8 to 2224.0] | 1817.8 [1194.5 to 2766.4] | 1585.6 [952.0 to 2640.9]
  Anti-HPV-16 Month 36 (N=28,12,11,9,16,15,15) | 1296.8 [917.1 to 1833.6] | 1200.5 [814.8 to 1768.9] | 1023.1 [389.2 to 2689.8] | 1275.3 [780.2 to 2084.7] | 960.6 [555.6 to 1660.7] | 1521.8 [943.4 to 2454.8] | 1076.9 [619.0 to 1873.6]
  Anti-HPV-16 Month 48 (N=28,12,11,9,16,15,15) | 1300.9 [952.3 to 1777.1] | 1115.4 [780.3 to 1594.3] | 1007.5 [361.3 to 2809.6] | 1337.7 [755.4 to 2368.9] | 1070.8 [614.6 to 1865.7] | 1417.8 [882.0 to 2279.0] | 1105.5 [620.6 to 1969.3]

3. Primary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus-16 (HPV-16) Antibodies
Description: Antibody titers were expressed as GMTs. The reference cut-off value was greater than or equal to (≥) 8 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 33 | 18 | 16 | 18 | 18 | 20 | 19
Titers
  Anti-HPV-16 Month 18 (N=32,15,13,16,16,17,17) | 1902.6 [1309.3 to 2764.7] | 1558.5 [1122.9 to 2163.2] | 1791.7 [823.6 to 3897.7] | 1552.9 [981.6 to 2456.5] | 1242.8 [687.3 to 2247.4] | 1869.6 [1161.1 to 3010.5] | 1764.4 [1073.8 to 2899.2]
  Anti-HPV-16 Month 24 (N=33,18,16,18,18,20,19) | 1472.8 [1046.2 to 2073.3] | 1223.4 [911.2 to 1642.6] | 1347.4 [740.7 to 2451.1] | 1579.5 [1053.9 to 2367.2] | 1092.8 [626.2 to 1907.2] | 1672.2 [1130.2 to 2474.1] | 1130.2 [1130.2 to 2367.2]
  Anti-HPV-16 Month 36 (N=33,18,16,18,18,20,19) | 1291.7 [928.4 to 1797.1] | 1031.2 [764.2 to 1391.5] | 1032.9 [538.9 to 1979.5] | 1107.7 [776.4 to 1580.3] | 841.4 [495.4 to 1428.9] | 1381.9 [901.0 to 2119.3] | 1128.6 [728.5 to 1748.3]
  Anti-HPV-16 Month 48 (N=33,18,16,18,18,20,19) | 1248.8 [907.1 to 1719.1] | 955.5 [722.7 to 1263.1] | 1104.9 [556.9 to 2192.1] | 1097.4 [737.8 to 1632.4] | 911.3 [526.5 to 1577.4] | 1310.1 [862.8 to 1989.2] | 1150.4 [727.8 to 1818.3]

4. Primary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus-18 (HPV-18) Antibodies.
Description: Seroconversion was defined as the appearance of antibodies in the serum of subjects seronegative before vaccination. Seronegative subjects are subjects who had an antibody concentration below cut-off value. The assessed cut-off value was 7 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 26 | 13 | 14 | 18 | 12 | 18 | 17
subjects
  Anti-HPV-18 Month 18 (N=26,10,12,16,11,15,15) | 26 | 10 | 12 | 16 | 11 | 15 | 15
  Anti-HPV-18 Month 24 (N=26,13,14,18,12,18,17) | 26 | 13 | 14 | 18 | 12 | 18 | 17
  Anti-HPV-18 Month 36 (N=26,13,14,18,12,18,17) | 26 | 13 | 14 | 18 | 12 | 18 | 17
  Anti-HPV-18 Month 48 (N=26,13,14,18,12,18,17) | 26 | 13 | 14 | 18 | 12 | 18 | 17

5. Primary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus-18 (HPV-18) Antibodies.
Description: Antibody titers were expressed as GMTs. The reference cut-off value was ≥ 7 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 26 | 13 | 14 | 18 | 12 | 18 | 17
EL.U/mL
  Anti-HPV-18 Month 18 (N=26,10,12,16,11,15,15) | 1060.9 [720.1 to 1562.9] | 469.3 [247.6 to 889.4] | 532.5 [211.2 to 1342.7] | 536.7 [296.0 to 973.0] | 563.7 [262.0 to 1212.5] | 637.9 [394.8 to 1030.8] | 572.2 [342.7 to 955.3]
  Anti-HPV-18 Month 24 (N=26,13,14,18,12,18,17) | 781.7 [538.5 to 1134.9] | 321.2 [192.8 to 535.2] | 387.0 [185.7 to 806.6] | 465.1 [267.6 to 808.5] | 502.4 [225.1 to 1121.5] | 536.5 [358.9 to 802.0] | 419.7 [269.1 to 654.5]
  Anti-HPV-18 Month 36 (N=26,13,14,18,12,18,17) | 733.6 [487.2 to 1104.6] | 286.1 [179.4 to 456.1] | 333.4 [151.0 to 736.0] | 424.6 [254.4 to 708.5] | 381.7 [165.1 to 882.7] | 456.5 [299.8 to 695.2] | 356.7 [232.3 to 547.8]
  Anti-HPV-18 Month 48 (N=26,13,14,18,12,18,17) | 729.3 [516.0 to 1030.8] | 248.6 [149.7 to 412.8] | 278.3 [125.6 to 616.6] | 443.3 [252.6 to 778.0] | 382.0 [170.8 to 854.0] | 440.7 [290.2 to 669.2] | 320.9 [206.2 to 499.2]

6. Primary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus-18 (HPV-18) Antibodies
Description: Antibody titers were expressed as GMTs. The reference cut-off value was greater than or equal to (≥) 7 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 33 | 18 | 16 | 18 | 18 | 20 | 19
Titers
  Anti-HPV-16 Month 18 (N=32,15,13,16,16,17,17) | 994.4 [699.5 to 1413.5] | 525.5 [328.2 to 841.6] | 524.1 [225.6 to 1217.5] | 536.7 [296.0 to 973.0] | 551.1 [312.4 to 972.2] | 574.9 [355.3 to 930.2] | 570.5 [365.6 to 890.4]
  Anti-HPV-16 Month 24 (N=33,18,16,18,18,20,19) | 739.5 [526.6 to 1038.3] | 355.2 [236.2 to 534.3] | 410.5 [217.0 to 776.6] | 465.1 [267.6 to 808.5] | 442.1 [251.9 to 775.8] | 497.7 [329.4 to 752.1] | 425.4 [287.1 to 630.5]
  Anti-HPV-16 Month 36 (N=33,18,16,18,18,20,19) | 683.5 [475.4 to 982.7] | 320.5 [220.4 to 466.1] | 349.8 [175.7 to 696.5] | 424.6 [254.4 to 708.5] | 348.1 [193.0 to 628.1] | 426.1 [281.7 to 644.4] | 364.9 [249.2 to 534.4]
  Anti-HPV-16 Month 48 (N=33,18,16,18,18,20,19) | 666.3 [477.9 to 929.2] | 284.6 [190.8 to 424.7] | 297.7 [148.9 to 595.3] | 443.3 [252.6 to 778.0] | 329.7 [184.8 to 588.2] | 412.0 [273.3 to 621.0] | 330.2 [222.3 to 490.4]

7. Secondary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus-31 (HPV-31) Antibodies.
Description: Seroconversion was defined as the appearance of antibodies in the serum of subjects seronegative before vaccination. Seronegative subjects are subjects who had an antibody concentration below cut-off value. The assessed cut-off value was 59 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 28 | 16 | 15 | 15 | 16 | 18 | 19
subjects
  Anti-HPV-31 Month 18 (N=27,13,12,13,14,15,17) | 25 | 13 | 12 | 13 | 14 | 15 | 17
  Anti-HPV-31 Month 24 (N=28,16,15,15,16,17,19) | 22 | 16 | 15 | 15 | 16 | 17 | 19
  Anti-HPV-31 Month 36 (N=28,16,15,15,16,18,19) | 23 | 16 | 15 | 15 | 16 | 18 | 19
  Anti-HPV-31 Month 48 (N=28,16,15,15,16,18,19) | 23 | 16 | 15 | 15 | 16 | 18 | 19

8. Secondary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus-31 (HPV-31) Antibodies.
Description: Antibody titers were expressed as GMTs. The reference cut-off value was ≥ 59 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL.
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 28 | 16 | 15 | 15 | 16 | 18 | 19
EL.U/mL.
  Anti-HPV-31 Month 18 (N=27,13,12,13,14,15,17) | 187.7 [124.2 to 283.8] | 1776.8 [1086.4 to 2906.1] | 2685.9 [1157.8 to 6230.9] | 2388.8 [1352.0 to 4220.8] | 2714.9 [1312.1 to 5617.3] | 1952.4 [1226.4 to 3108.2] | 3466.4 [2077.8 to 5782.9]
  Anti-HPV-31 Month 24 (N=28,16,15,15,16,17,19) | 125.3 [80.6 to 194.8] | 1336.1 [891.6 to 2002.2] | 2076.2 [1168.0 to 3690.7] | 1966.7 [1221.9 to 3165.5] | 2298.0 [1214.8 to 4347.0] | 1911.8 [1162.0 to 3145.5] | 2518.3 [1648.7 to 3846.7]
  Anti-HPV-31 Month 36 (N=28,16,15,15,16,18,19) | 164.6 [107.7 to 251.7] | 1346.7 [941.1 to 1927.0] | 1776.6 [976.5 to 3232.1] | 1644.0 [993.6 to 2720.2] | 1825.1 [984.1 to 3384.7] | 1584.1 [982.1 to 2555.2] | 2080.0 [1400.9 to 3088.3]
  Anti-HPV-31 Month 48 (N=28,16,15,15,16,18,19) | 174.7 [114.4 to 266.7] | 1284.5 [878.4 to 1878.3] | 2105.3 [1155.1 to 3837.3] | 1744.2 [966.3 to 3148.3] | 2126.9 [1159.6 to 3901.1] | 1434.2 [892.0 to 2306.0] | 2118.1 [1536.6 to 2919.7]

9. Secondary Outcome: Number of Seroconverted Subjects Against Human Papillomavirus-45 (HPV-45) Antibodies.
Description: as for outcome 7
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 24 | 17 | 12 | 13 | 16 | 18 | 16
subjects
  Anti-HPV-45 Month 18 (N=20,14,10,11,14,15,15) | 20 | 14 | 10 | 11 | 14 | 15 | 15
  Anti-HPV-45 Month 24 (N=19,17,12,13,16,17,16) | 19 | 17 | 12 | 13 | 16 | 17 | 16
  Anti-HPV-45 Month 36 (N=18,17,12,13,16,18,16) | 18 | 17 | 12 | 13 | 16 | 18 | 16
  Anti-HPV-45 Month 48 (N=19,17,12,13,16,18,16) | 19 | 17 | 12 | 13 | 16 | 18 | 16

10. Secondary Outcome: Geometric Mean Titers (GMTs) for Human Papillomavirus-45 (HPV-45) Antibodies.
Description: Antibody titers were expressed as GMTs. The reference cut-off value was ≥ 59 EL.U/mL.
Time Frame: At Months 18, 24, 36 and 48.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 24 | 17 | 12 | 13 | 16 | 18 | 16
EL.U/mL
  Anti-HPV-45 Month 18 (N=20,14,10,11,14,15,15) | 184.8 [111.9 to 305.1] | 919.8 [510.9 to 1655.9] | 1731.0 [591.8 to 5063.3] | 959.1 [557.9 to 1648.9] | 1086.6 [528.7 to 2233.2] | 1235.8 [757.9 to 2014.8] | 1094.9 [613.1 to 1955.4]
  Anti-HPV-45 Month 24 (N=19,17,12,13,16,17,16) | 138.3 [86.4 to 221.4] | 713.0 [440.6 to 1153.9] | 1274.5 [590.1 to 2752.5] | 904.9 [546.7 to 1497.8] | 948.1 [515.2 to 1744.6] | 1106.5 [680.1 to 1800.4] | 848.2 [494.1 to 1456.0]
  Anti-HPV-45 Month 36 (N=18,17,12,13,16,18,16) | 165.4 [97.9 to 279.4] | 707.8 [451.9 to 1108.6] | 1103.9 [521.0 to 2338.8] | 810.7 [492.6 to 1334.2] | 825.2 [450.2 to 1512.4] | 1015.6 [660.2 to 1562.4] | 774.7 [486.2 to 1234.3]
  Anti-HPV-45 Month 48 (N=19,17,12,13,16,18,16) | 190.7 [115.8 to 314.1] | 659.0 [415.4 to 1045.6] | 1036.2 [477.2 to 2249.9] | 806.9 [447.5 to 1454.7] | 815.1 [453.3 to 1465.7] | 914.6 [600.7 to 1392.5] | 750.0 [448.0 to 1255.5]

11. Secondary Outcome: Number of Subjects With at Least One New Onset of Chronic Disease (NOCDs)
Description: NOCDs include conditions such as diabetes, autoimmune disease, asthma, allergies etc. At least one NOCD = At least one NOCD experienced (regardless of the Medical Dictionary for Regulatory Activities [MedDRA] Preferred Term)
Time Frame: From Month 0 to Months 18, 24, 36 and 48
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  NOCD(s) at Month 18 | 6 | 1 | 6 | 2 | 3 | 1 | 2
  NOCD(s) at Month 24 | 6 | 1 | 6 | 2 | 3 | 1 | 2
  NOCD(s) at Month 36 | 7 | 1 | 6 | 2 | 3 | 1 | 3
  NOCD(s) at Month 48 | 7 | 1 | 7 | 3 | 4 | 1 | 4

12. Secondary Outcome: Number of Subjects With at Least One Medically Significant Condition (MAEs).
Description: MAEs were defined as adverse events (AEs) prompting emergency room or physician visits that were not related to common diseases or routine visits for physical examination or vaccination, or serious adverse events (SAEs) that were not related to common diseases. Common diseases included: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities, and injury. At least one MAE = At least one medically significant AE experienced (regardless of the MedDRA Preferred Term).
Time Frame: From Month 0 to Months 18, 24, 36 and 48
Population: as for outcome 11
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  MAE(s) at Month 18 | 4 | 3 | 2 | 4 | 5 | 1 | 1
  MAE(s) at Month 24 | 6 | 3 | 3 | 7 | 8 | 5 | 1
  MAE(s) at Month 36 | 9 | 4 | 3 | 7 | 9 | 5 | 2
  MAE(s) at Month 48 | 14 | 7 | 5 | 9 | 12 | 5 | 3

13. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity, or are a congenital anomaly/birth defect in the offspring of a study subject. Any = Occurrence of any symptom regardless of intensity grade.
Time Frame: From Month 0 to Months 18, 24, 36 and 48
Population: as for outcome 11
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  Any SAE(s) at Month 18 | 2 | 3 | 1 | 3 | 2 | 0 | 1
  Any SAE(s) at Month 24 | 2 | 3 | 1 | 3 | 3 | 1 | 1
  Any SAE(s) at Month 36 | 2 | 3 | 2 | 4 | 3 | 1 | 1
  Any SAE(s) at Month 48 | 6 | 4 | 2 | 6 | 3 | 1 | 1

14. Secondary Outcome: Number of Subjects With Pregnancy Outcomes.
Description: Pregnancy outcomes were healthy baby, spontaneous abortion and elective abortion.
Time Frame: From Month 0 to Month 18
Population: as for outcome 11
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  Healthy baby | 3 | 0 | 2 | 1 | 0 | 1 | 3
  Spontaneous abortion | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Elective abortion | 1 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With Pregnancy Outcomes.
Description: Pregnancy outcomes were healthy baby, spontaneous abortion, elective abortion and ongoing pregnancy.
Time Frame: From Month 0 to Month 24
Population: as for outcome 11
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  Healthy baby | 4 | 1 | 2 | 2 | 0 | 1 | 3
  Spontaneous abortion | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Elective abortion | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Ongoing pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Pregnancy Outcomes.
Description: Pregnancy outcomes were healthy baby, abnormal infant/congenital anomaly, spontaneous abortion and elective abortion.
Time Frame: From Month 0 to Month 36
Population: as for outcome 11
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  Healthy baby | 4 | 4 | 3 | 2 | 0 | 1 | 3
  Abnormal infant/congenital anomaly | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Spontaneous abortion | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Elective abortion | 1 | 0 | 0 | 1 | 0 | 0 | 0

17. Secondary Outcome: Number of Subjects With Pregnancy Outcomes.
Description: Pregnancy outcomes were normal infant, abnormal infant/congenital anomaly, spontaneous abortion and elective termination.
Time Frame: From Month 0 to Month 48
Population: as for outcome 11
Measure: Number; unit: subjects
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
subjects
  Normal infant | 9 | 6 | 3 | 2 | 0 | 1 | 4
  Abnormal infant/congenital anomaly | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Spontaneous abortion | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Elective termination | 1 | 0 | 0 | 1 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: SAE(s): during the entire study period (i.e. Months 0-48); No Unsolicited AE(s) and solicited local/general symptoms data were collected during this study.
Arm/Group | Cervarix Group | Cervarix 1 Group | Cervarix 2 Group | Cervarix 3 Group | Cervarix 4 Group | Cervarix 5 Group | Cervarix 6 Group
Serious Adverse Events (participants affected / at risk) | 6/88 | 4/50 | 2/49 | 6/48 | 3/48 | 1/50 | 1/50
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=88) | Cervarix 1 Group (N=50) | Cervarix 2 Group (N=49) | Cervarix 3 Group (N=48) | Cervarix 4 Group (N=48) | Cervarix 5 Group (N=50) | Cervarix 6 Group (N=50)
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myelitis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bulimia nervosa (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.